CLINICAL TRIAL: NCT03667209
Title: Exercise and Pain Neuroscience Education for Patients With Neck Pain: Impact
Brief Title: Exercise and Pain Neuroscience Education for Patients With Neck Pain: Impact on Pain and Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21/2018
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2018-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional exercise and pain neuroscience education (Experimental): Will include exercises of the neck and scapular regions using traditional methods and pain neuroscience education
  Interventions: Other: Pain neuroscience education (PNE) and traditional exercise
- Suspension exercise and pain neuroscience education (Active Comparator): Will include suspension exercises of the neck and scapular regions using traditional methods and pain education.
  Interventions: Other: Pain neuroscience education (PNE) and suspension exercise

INTERVENTIONS:
Other: Pain neuroscience education (PNE) and traditional exercise — PNE will cover the neurophysiology of pain, transition from acute to chronic pain and the nervous system ability to modulate the pain experience.
  Exercise of the neck and scapular regions, including strength, motor control and stretching exercises.
  Initially (first 3 sessions) will be delivered individually and then (last 3 sessions)in small groups (4 participants). A total of 6 sessions will be delivered during 6 weeks. Each session will take around 1 hour.
  Arms: Traditional exercise and pain neuroscience education
Other: Pain neuroscience education (PNE) and suspension exercise — PNE will cover the neurophysiology of pain, transition from acute to chronic pain and the nervous system ability to modulate the pain experience.
  Exercise of the neck and scapular regions, including strength, motor control and stretching exercises. delivered in suspension.
  Initially (first 3 sessions) will be delivered individually and then (last 3 sessions)in small groups (4 participants). A total of 6 sessions will be delivered during 6 weeks. Each session will take around 1 hour.
  Arms: Suspension exercise and pain neuroscience education

SUMMARY:
This study will compare the effectiveness of pain neuroscience education and neck/shoulder traditional exercises versus pain neuroscience education and neck/shoulder suspension training exercises for patients with chronic idiopathic neck pain (CINP).

DETAILED DESCRIPTION:
The investigators anticipate that 66 patients with chronic idiopathic neck pain will be randomized to receive pain neuroscience education and shoulder/neck traditional exercises (n=33) or pain neuroscience education and shoulder/neck suspension exercises (n=33). Data on pain intensity (Visual Analogue Scale), pain disability, neck flexor and extensor muscles endurance, scapulae stabilizers endurance, pain catastrophizing (Pain catastrophizing Scale), trait and state anxiety (State-Trait Anxiety Inventory) and knowledge of pain neurophysiology (Neurophysiology of Pain Questionnaire) will be collected. Measurements will be taken before, after the intervention and at 3 months follow up.

Statistical analysis will be performed using a mixed-methods ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic idiopathic neck pain.

Exclusion Criteria:

* Cervical radiculopathy
* Neck fractures
* Tumors
* Rheumatological disorders
* Any other serious cause of neck pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: VAS | Baseline
  Method of assessment - Visual analogue scale (VAS), which measures pain intensity from a minimum of 0 to a maximum of 10 (maximum pain intensity).
Pain intensity: VAS | 7 weeks
  Method of assessment - Visual analogue scale (VAS), which measures pain intensity from a minimum of 0 to a maximum of 10 (maximum pain intensity).
Pain intensity: VAS | 6 months
  Method of assessment - Visual analogue scale (VAS), which measures pain intensity from a minimum of 0 to a maximum of 10 (maximum pain intensity).
Neck pain associated disability | Baseline
  Method of assessment - the Neck Disability Index, which is a disability index with 5 questions on neck pain associated disability that ranges from 0 (no disability) to 50 (complete disability).
Neck pain associated disability | 7 weeks
  Method of assessment - the Neck Disability Index, which is a disability index with 5 questions on neck pain associated disability that ranges from 0 (no disability) to 50 (complete disability).
Neck pain associated disability | 6 months
  Method of assessment - the Neck Disability Index, which is a disability index with 5 questions on neck pain associated disability that ranges from 0 (no disability) to 50 (complete disability).

SECONDARY OUTCOMES:
Neck pain frequency | Baseline
  Method of assessment - a question on neck pain frequency in the previous week (never, seldom, occasionally, often, always)
Neck pain frequency | 7 weeks
  Method of assessment - a question on neck pain frequency in the previous week (never, seldom, occasionally, often, always)
Neck pain frequency | 6 months
  Method of assessment - a question on neck pain frequency in the previous week (never, seldom, occasionally, often, always)
Neck pain location | Baseline
  Method of assessment - a body chart where the patients will draw where he/she feels pain
Neck pain location | 7 weeks
  Method of assessment - a body chart where the patients will draw where he/she feels pain
Neck pain location | 6 months
  Method of assessment - a body chart where the patients will draw where he/she feels pain
Neck flexor muscles endurance test | Baseline
  Method of assessment - physical test; the participant is in supine and he/she is asked to flex the upper cervical spine, move their head away from the couch approximately 2.5 cm and then maintain this position for as long as possible. The test result is the time (in seconds) that each participant holds the position.
Neck flexor muscles endurance test | 7 weeks
  Method of assessment - physical test; the participant is in supine and he/she is asked to flex the upper cervical spine, move their head away from the couch approximately 2.5 cm and then maintain this position for as long as possible. The test result is the time (in seconds) that each participant holds the position.
Neck flexor muscles endurance test | 6 months
  Method of assessment - physical test; the participant is in supine and he/she is asked to flex the upper cervical spine, move their head away from the couch approximately 2.5 cm and then maintain this position for as long as possible. The test result is the time (in seconds) that each participant holds the position.
Neck extensor muscles endurance test | Baseline
  Method of assessment - physical test; the participant is in prone and position, head neutral, and supporting 2 Kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining the neutral head positioning. The test result is the time (in seconds) that each participant holds the position.
Neck extensor muscles endurance test | 7 weeks
  Method of assessment - physical test; the participant is in prone and position, head neutral, and supporting 2 Kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining the neutral head positioning. The test result is the time (in seconds) that each participant holds the position.
Neck extensor muscles endurance test | 6 months
  Method of assessment - physical test; the participant is in prone and position, head neutral, and supporting 2 Kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining the neutral head positioning. The test result is the time (in seconds) that each participant holds the position.
Scapular stabilizers' endurance test | Baseline
  Method of assessment - physical test; Participants were standing with the shoulders and elbows flexed at 90º, while pulling both extremities of a dynamometer to reach 1 Kg of force. The test result is the time (in seconds) that each participants was able to hold this position.
Scapular stabilizers' endurance test | 7 weeks
  Method of assessment - physical test; Participants were standing with the shoulders and elbows flexed at 90º, while pulling both extremities of a dynamometer to reach 1 Kg of force. The test result is the time (in seconds) that each participants was able to hold this position.
Scapular stabilizers' endurance test | 6 months
  Method of assessment - physical test; Participants were standing with the shoulders and elbows flexed at 90º, while pulling both extremities of a dynamometer to reach 1 Kg of force. The test result is the time (in seconds) that each participants was able to hold this position.
Pain Catastrophizing Scale | Baseline
  Method of assessment - the Pain Catastrophizing Scale; score ranges from 0 (no catastrophizing) to 52 (maximum catastrophizing).
Pain Catastrophizing Scale | 7 weeks
  Method of assessment - the Pain Catastrophizing Scale; score ranges from 0 (no catastrophizing) to 52 (maximum catastrophizing).
Pain Catastrophizing Scale | 6 months
  Method of assessment - the Pain Catastrophizing Scale; score ranges from 0 (no catastrophizing) to 52 (maximum catastrophizing).
Neurophysiology of pain questionnaire | Baseline
  Method of assessment - the Neurophysiology of pain questionnaire which measures the patients' knowledge on pain neurophysiology; score ranges from 0 to 19 and the higher the score the more patients know on pain neurophysiology.
Neurophysiology of pain questionnaire | 7 weeks
  Method of assessment - the Neurophysiology of pain questionnaire which measures the patients' knowledge on pain neurophysiology; score ranges from 0 to 19 and the higher the score the more patients know on pain neurophysiology.
Neurophysiology of pain questionnaire | 6 months
  Method of assessment - the Neurophysiology of pain questionnaire which measures the patients' knowledge on pain neurophysiology; score ranges from 0 to 19 and the higher the score the more patients know on pain neurophysiology.
Patients' Global Impression of Change | Baseline
  Method of assessment - the Patients' Global Impression of Change is a 7 point numeric rating scale; a score of 5 or more in the PGIC is associated with a clinically significant improvement in the patients' condition.
Patients' Global Impression of Change | 7 weeks
  Method of assessment - the Patients' Global Impression of Change is a 7 point numeric rating scale; a score of 5 or more in the PGIC is associated with a clinically significant improvement in the patients' condition.
Patients' Global Impression of Change | 6 months
  Method of assessment - the Patients' Global Impression of Change is a 7 point numeric rating scale; a score of 5 or more in the PGIC is associated with a clinically significant improvement in the patients' condition.
TAMPA scale of kinesiophobia | Baseline
  Method of assessment - the TAMPA scale of kinesiophobia assesses fear of movement and its score ranges from 13 to 52; the higher the score the higher the fear of movement.
TAMPA scale of kinesiophobia | 7 weeks
  Method of assessment - the TAMPA scale of kinesiophobia assesses fear of movement and its score ranges from 13 to 52; the higher the score the higher the fear of movement.
TAMPA scale of kinesiophobia | 6 months
  Method of assessment - the TAMPA scale of kinesiophobia assesses fear of movement and its score ranges from 13 to 52; the higher the score the higher the fear of movement.
Chronic Pain Coping Inventory | Baseline
  Method of assessment - Chronic Pain Coping Inventory is a scale that assesses patient coping strategies; Patients are asked to rate the number of days (0-7 days) over the past week when they used each of 65 strategies at least once.
Chronic Pain Coping Inventory | 7 weeks
  Method of assessment - Chronic Pain Coping Inventory is a scale that assesses patient coping strategies; Patients are asked to rate the number of days (0-7 days) over the past week when they used each of 65 strategies at least once.
Chronic Pain Coping Inventory | 6 months
  Method of assessment - Chronic Pain Coping Inventory is a scale that assesses patient coping strategies; Patients are asked to rate the number of days (0-7 days) over the past week when they used each of 65 strategies at least once.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No